CLINICAL TRIAL: NCT00239031
Title: Multicentre, Controlled, Prospective, Randomized, Open-label Clinical Trial to Compare Enteric-Coated Mycophenolate Sodium (EC-MPS) Plus Reduced Dose Cyclosporine Microemulsion (CsA-ME) Vs EC-MPS Plus Standard Dose CsA-ME in Elderly de Novo Renal Transplant Recipients Treated With Basiliximab and Short-term Steroids
Brief Title: Study of Enteric-Coated Mycophenolate Sodium (EC-MPS) Plus Reduced-dose Cyclosporine Microemulsion (CsA-ME) Compared to EC-MPS Plus Standard Dose CsA-ME in Eldery de Novo Renal Transplant Recipients Treated With Basiliximab and Short-term Steroids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CERL080A2405IT01
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Denovo Renal Transplantation
Keywords: Renal transplantation, EC-MPS

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Enteric-Coated Mycophenolate Sodium

INTERVENTIONS:
Drug: Enteric-Coated Mycophenolate Sodium — Enteric-Coated Mycophenolate Sodium

SUMMARY:
All patients of the core study who are interested of being treated with EC-MPS will be included in an open-label extension study to collect further information on the long-term safety, tolerability and efficacy of this drug.

The aim of this study is to compare the renal function, 6 months after transplant, in de novo old-age renal transplant recipients treated with EC-MPS plus reduced dose CsA-ME or with EC-MPS plus standard dose CsA-ME, both in combination with basiliximab and short-term oral steroids.

ELIGIBILITY:
Inclusion criteria Male or female patients 55_75 years old, recipients of a primary kidney transplant from a cadaver donor Subjects in whom CsA-ME plus basiliximab is selected as basic immunosuppressive regimen.

Cold ischemia time 20 hrs. Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to enrollment and must use an effective contraception during the trial and for 6 weeks following discontinuation of the study medication.

Patients who are willing and able to participate in the full course of the study and from whom written informed consent has been obtained.

Exclusion criteria Multi-organ recipients (e.g. kidney and pancreas, double kidney) or any previous transplant.

Patients with any known hypersensitivity to mycophenolic acid or other components of the formulation (e.g. lactose).

Patients with thrombocytopenia (75,000 mm), with an absolute neutrophil count of 1,500 mm and or leukocytopenia ( 2,500 mm3) and/or hemoglobin < 6 g/dL at Screening or Baseline.

Patients who have received an investigational drug within four weeks prior to study entry.

Patients with a history of malignancy within the last five years, except excised squamous or basal cell carcinoma of the skin.

Females of childbearing potential who are planning to become pregnant, who are pregnant and or lactating, who are unwilling to use effective means of contraception.

Presence of clinically significant infections requiring continued therapy. Known positivity to HIV or positive HBsAg test. Evidence of drug and or alcohol abuse Existence of any surgical or medical condition, other than the current transplant, which in the opinion of the investigator might significantly alter the absorption, distribution, metabolism or excretion of study medication, and/or presence of severe diarrhea, active peptic ulcer disease, or uncontrolled diabetes mellitus.

Patients with Panel Reactive Antibodies (PRA) historical peak evaluation 30% or most recent evaluation 15%.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2002-03; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
The 6-month study values of creatinine clearance, as calculated according to Cockcroft and Gault, summarized and compared between treatment groups.

SECONDARY OUTCOMES:
Incidence of treatment failure (biopsy-proven and/or treated acute rejection, graft loss, death or loss to follow-up at 6 and 12 months;
Incidence of biopsy proven acute rejection at Month 6 and 12
Incidence of graft loss at Month 6 and 12
Rate of delayed graft function (DGF) and the time to adequate renal function (serum creatinine < 2,5 mg/dL);
Pharmacokinetics of MPA and MPAG at Day 15, Month 3 and Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis